CLINICAL TRIAL: NCT06276296
Title: Evaluation of Heart Rate Variability in Patients After Ablation Using Pulsed Field and Radiofrequency
Brief Title: Heart Rate Variability After Ablation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Vascular surgery, University hospital Královské Vinohrady, Prague (Other)
Responsible Party: Sponsor
Other Study IDs: 0001
Record Dates: First submitted 2024-02-06; First posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Heart rate variability; Pulsed field ablation; Radiofrequency ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electrocardiography, Ambulatory; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PFA group: Patients undergoing pulsed field ablation
  Interventions: Diagnostic Test: Holter EKG - 1 day before ablation; Procedure: Pulsed field ablation; Diagnostic Test: Holter EKG - 1 month after ablation
- RFA group: Patients undergoing radiofrequency ablation
  Interventions: Diagnostic Test: Holter EKG - 1 day before ablation; Procedure: Radiofrequency ablation; Diagnostic Test: Holter EKG - 1 month after ablation

INTERVENTIONS:
Diagnostic Test: Holter EKG - 1 day before ablation — 24 hours Holter EKG - 1 day before ablation
Procedure: Radiofrequency ablation — Pulmonary vein isolation using radiofrequency ablation
  Groups: RFA group
Procedure: Pulsed field ablation — Pulmonary vein isolation using pulsed field ablation
  Groups: PFA group
Diagnostic Test: Holter EKG - 1 month after ablation — 24 hours Holter EKG 1 month after ablation

SUMMARY:
Pulsed-field catheter ablation is a promising new treatment method for patients with atrial fibrillation. The mechanism of cell damage here is different from that of classic catheter ablation, in which the ganglion plexuses around the pulmonary veins are also damaged and thus changes in the autonomic nervous system occur. The aim of the work is to find out, using heart rate variability, whether the autonomic system is less affected during pulsed field ablation than in classic radiofrequency ablation.

DETAILED DESCRIPTION:
Catheter ablation for pulmonary vein isolation (PVI) is the most effective treatment method for atrial fibrillation (AF). For a long time, radiofrequency energy (RFA) was dominantly used for ablation, which leads to tissue heating and thus thermal damage. The methodology of pulsed-field ablation, or irreversible electroporation, has been completely newly developed. This form of energy does not lead to thermal tissue damage (as is the case with radiofrequency energy), but with the help of high-intensity nanopulses of electrical energy, the ion channels of cardiomyocytes are permanently opened, the concentration gradient of ions is canceled and thus their irreversible destruction. In addition to the electrical isolation of the pulmonary vein, standard radiofrequency isolation of the pulmonary veins leads to the ablation of collateral ganglion plexuses and thus to the influence of the autonomic nervous system. This is very positive, an imbalance between sympathetic and parasympathetic innervating the left atrium is considered a risk factor for AF induction, and its damage with standard RFA is considered part of the RFA ablation effect. Available studies suggest that PFA probably induces significantly weaker and less permanent suppression of cardiac autonomic regulation compared to RF energy used for PVI.

Measuring heart rate variability is a simple non-invasive method. A regular ECG Holter recorder can be used for the measurement. Patients will be fitted with a 24-hour Holter ECG on admission to determine the original heart rate variability. Catheter ablation will take place the next day. Patients will be treated using one of two methods of pulmonary vein isolation - RFA or PFA. One month after the catheterization procedure, a 24-hour Holter ECG will be used again to detect changes in HRV compared to preoperative values.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal atrial fibrillation
* indication for catheter ablation due to atrial fibrillation
* willingness to participate

Exclusion Criteria:

* atrial fibrillation throughout Holter ECG recording
* significant valve disease
* left ventricular dysfunction, EF less than 35%

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with paroxysmal symptomatic atrial fibrillation fulfilling standard criteria for catheter ablation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Mean RR interval (ms) | 1 month
  Time domain parameter
SDNN (ms) | 1 month
  Standard deviation of RR intervals - time domain parameter
RMSSD (ms) | 1 month
  root mean square of successive differences - time domain parameter
pNN50 (%) | 1 month
  the number of successive intervals differing more than 50 ms or the corresponding relative amount - time domain parameter
peak frequency (Hz) | 1 month
  The frequency-domain measures extracted from a spectrum estimate for each frequency band (very low, low and high)
power (ms2) | 1 month
  A parameter obtained from the estimation of the frequency spectrum
LF/HF ratio | 1 month
  Ratio between low frequency and high frequency band powers
SD1 (ms) | 1 month
  In Poincaré plot, the standard deviation perpendicular to the line-of-identity
SD2 (ms) | 1 month
  In Poincaré plot, the standard deviation along the line-of-identity
SD2/SD1 | 1 month
  Ratio between SD2 and SD1
ApEn | 1 month
  Approximate entropy
Correlation dimension | 1 month
  The correlation dimension is expected to give information on the minimum number of dynamic variables needed to model the underlying system

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiocenter, 3rd Medical School, Charles University and University Hospital Kralovske Vinohrady, Prague, Czechia